CLINICAL TRIAL: NCT06006455
Title: An Evaluation of the Effect of the Erchonia® LunulaLaser™ for the Treatment of Toenail Onychomycosis
Brief Title: Effect of the Erchonia® LunulaLaser™ for the Treatment of Toenail Onychomycosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated early by the sponsor for business reasons unrelated to safety. No data analysis was performed.
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-TOT
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Results first posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Onychomycosis of Toenail

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Erchonia LunulaLaser (Experimental): The Erchonia LunulaLaser emits red light (635 nm) and violet light (405 nm) to the affected toenail for 12 minutes per treatment. The treatment phase involves an initial weekly treatment administration phase, 1 treatment a week for 4 weeks, followed by an every two-month maintenance treatment administration phase, months 3, 5, 7, 9, and 11.
  Interventions: Device: Erchonia LunulaLaser

INTERVENTIONS:
Device: Erchonia LunulaLaser — 405nm violet and 635nm red laser light therapy.

SUMMARY:
The purpose of this clinical study is to demonstrate the efficacy of the Erchonia LunulaLaser™, for the treatment of onychomycosis of the toenail.

DETAILED DESCRIPTION:
This active test treatment group only study will evaluate the effectiveness of the Erchonia LunulaLaser™ manufactured by Erchonia Corporation (the Sponsor) for the treatment of onychomycosis of the toenail.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of the presence of fungal infection through a positive KOH stain finding and a positive fungal culture finding
* Identification through fungal culture of the growth of Trichophyton rubrum (T. rubrum) or other common dermatophyte
* Visual clinical presentation of onychomycosis in the target great toenail is distal subungual onychomycosis (DSO), visualized as a nail with normal surface texture and thickness but variable "bays" of white nail that extend from the distal nail tip proximally into the area of the nail bed
* Clinical involvement of onychomycosis in the target toenail is between 20%-50%
* Subject is willing and able to refrain from employing other (non-study) treatments (traditional or alternative) for his or her toenail onychomycosis throughout study participation.
* Subject is willing and able to refrain from the use of nail cosmetics such as clear and/or colored nail lacquers throughout study participation
* Male or female
* 18 years of age or older

Exclusion Criteria:

* Lack of confirmation of the presence of fungal infection through a negative KOH stain finding and/or a negative fungal culture finding
* Visual clinical presentations of onychomycosis in the target great toenail that are inconsistent with the clinical presentation of distal subungual onychomycosis (DSO), in whole or in part (i.e. indicative of mixed etiology); specifically visual clinical presentations consistent with one or more of the following:

  * Proximal subungual onychomycosis (PSO): visualized as a white discoloration below the nail plate at the base of the nail, near the lunula. The distal nail retains normal appearance and texture. PSO involves infection near the matrix, deep to the nail. It may be associated with trauma to the nail or to immune compromise
  * Superficial white onychomycosis (SWO): visualized by the appearance of a white coating on the nail surface that can be eliminated by filing or buffing the surface of the affected portion of the nail
  * Complete dystrophy: Nails which are 100% dystrophic are manifested by yellowing and thickening of the entire nail unit
  * Other nail changes: Nails that visually present with changes that appear as parallel lines, small pinpoint depressions, brown spots, black or brown linear streaks, complete yellowing of all nails without textural change, green debris below the nail, or notches in the nail margin
* Less than 2mm clear (unaffected) nail plate length beyond the proximal fold
* Presence of dermatophytoma (thick masses of fungal hyphae and necrotic keratin between the nail plate and nail bed)
* Infection involving lunula e.g., genetic nail disorders, primentary disorders
* Severe plantar (moccasin) tinea pedis
* Psoriasis of the skin and/or nails, lichen planus, or other medical conditions known to induce nail changes
* Onychogryphosis
* Trauma from ill-fitting shoes, running, or overly-aggressive nail care
* Previous toenail surgery
* Uncontrolled diabetes mellitus
* Peripheral vascular disease
* Recurrent cellulitis
* Lymphatic insufficiency
* Immune compromise (whether due to underlying medical disorders or immunosuppressive treatments)
* Other compromised states of health
* Known photosensitivity disorder
* Use of oral antifungal drugs in the prior 6 months
* Use of topical treatment of the skin or nails within the prior 2 months
* Any abnormality of the toenail that could prevent a normal appearing nail from occurring if clearing of infection is achieved.
* Current trauma, open wound on or about the treatment area
* Deformity of the target toe/toenail secondary to fungal infection/onychomycosis due to prior injury, surgical procedures or another medical condition
* Pregnant or planning pregnancy prior to the end of study participation
* Serious mental health illness such as dementia or schizophrenia; psychiatric hospitalization in the past two years
* Developmental disability or cognitive impairment that would preclude adequate comprehension of the informed consent form and/or ability to follow study subject requirements and/or record the necessary study measurements
* Involvement in litigation and/or receiving disability benefits related in any way to the parameters of the study
* Participation in a clinical study or other type of research in the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin Stones, MB.ChB, Principal Investigator — Blemish Clinic
Locations (1):
- Blemish Clinic, Edenfield, Cheshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erchonia LunulaLaser
Started | 28
Completed | 25
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Erchonia LunulaLaser
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.32 (92.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 27
  Asian/ Pacific Islander | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Toenails Attaining Complete Cure
Description: Complete Cure criteria is defined as a subject/toenail satisfying both the 'Clinical Cure' and the 'Mycological Cure' criteria in order to be considered a study responder, defined as follows:
  (i) Clinical Cure: Measurement of clear nail increase as the following:
  * at least 12 mm increase in clear nail of the great toenail, with evidence of distal growth of the affected area, 12 months after the first treatment; or
  * complete clearance 12 months after the first treatment if less than 12 mm distal nail was involved prior to treatment.
  The response should be progressive in at least 2 sequential timepoints that are at least 3 months apart, with projected increase of at least 1 mm per month.
  (ii) Mycologic Cure: both negative KOH and negative Fungal Culture results (or two serial negative Fungal Culture results)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Erchonia LunulaLaser
Number analyzed (Participants) | 25
Participants | 6

2. Secondary Outcome: Mycologic Cure
Description: Mycological cure is defined as negative culture for dermatophytes using the BioMed InTray™ DM Culture
Time Frame: 14 months
Measure: Count of Participants; unit: Participants
Arm/Group | Erchonia LunulaLaser
Number analyzed (Participants) | 25
Participants | 14

ADVERSE EVENTS:
Time Frame: 14 months
Arm/Group | Erchonia LunulaLaser
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-06-20): https://cdn.clinicaltrials.gov/large-docs/55/NCT06006455/Prot_SAP_ICF_000.pdf